CLINICAL TRIAL: NCT06677307
Title: A Phase 1/2a, Single- and Multiple-dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of KRRO 110 in Healthy Adult Volunteers and in Adult Participants With Alpha-1 Antitrypsin Deficiency (AATD) (REWRITE)
Brief Title: A Phase 1/2a, Single- and Multiple-dose Escalation Study of KRRO-110
Acronym: REWRITE
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Korro Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KRRO-110-001
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Alpha-1 Anti-trypsin Deficiency; AATD
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: KRRO-110 (Part A and Part B) (Experimental): KRRO-110 is an RNA editing oligonucleotide encapsulated in a lipid nanoparticle (LNP) administered by intravenous (IV) infusion as a single dose in Part A (SAD), multi-dose in Part B (MAD).
  Interventions: Drug: KRRO-110
- Arm 2: Placebo (Part A only) (Placebo Comparator): Placebo, IV administration
  Interventions: Drug: KRRO-110

INTERVENTIONS:
Drug: KRRO-110 — KRRO-110 drug product, IV

SUMMARY:
The purpose of this first-in human (FIH) study is to assess the safety, tolerability, and pharmacokinetics (PK) of single and multiple doses of KRRO-110 in both healthy adult participants and in clinically stable patients with Alpha-1 antitrypsin deficiency (AATD).

ELIGIBILITY:
Inclusion Criteria:

Part A SAD cohort Inclusion Criteria (Healthy Volunteers)

* Adult male or female participants, 18 to 65 years of age
* Documented PiMM genotype
* Participants who are willing to and able to provide signed written informed consent

PiZZ Genotype (Part A SAD and Part B MAD cohorts) Inclusion Criteria (PiZZ Genotype)

* Adult male or female participants 18 to 70 years of age (inclusive)
* Documented PiZZ genotype
* Baseline blood total AAT level < 11 µM/L

Exclusion Criteria:

Exclusion Criteria (Healthy Volunteers)

* Female participant of childbearing potential or male participant that is unable or unwilling to use an approved, reliable means of contraception
* Body mass index (BMI) > 32 or < 18.5 kg/m2
* History or current clinical evidence of hepatic disease
* Evidence of active infection
* History of medical condition(s), eg, advance cardiac disease, current or recent malignancy, organ transplantation, or other illness
* Serology result indicative of any exposure (past or active) to hepatitis C, hepatitis B, or human immunodeficiency virus (HIV)
* Respiratory or other acute illness within 8 weeks
* Tobacco use of any kind within 6 months

Exclusion Criteria (PiZZ Genotype)

* Female participant of childbearing potential or male participant that is unable or unwilling to use an approved, reliable means of contraception
* BMI > 32 or < 18.5 kg/m2 or weight > 90 kg
* History of FEV1 < 35%
* History or current clinical evidence of advanced hepatic disease and/or pulmonary disease
* Use of an experimental therapy except KRRO-110 within 6 months or 5 half-lives for the experimental therapy, whichever is greater
* Tobacco use of any kind within 6 months
* Use of conventionally dosed AAT augmentation therapy within 5 half-lives
* Serology result consistent with exposure to HIV, or serology consistent with active hepatitis B or hepatitis C infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | From Day 1 to Day 43 in the SAD and from Day 1 to Day 85 in the MAD
  Type, frequency, and severity of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of KRRO-110 | Day 1 to Day 43 (SAD), and Day 1 to Day 85 (MAD)
  PK profile of KRRO-110 including maximum blood concentration (Cmax)
Pharmacodynamics (PD) of KRRO-110 | Day 1 to Day 43 (SAD), and Day 1 to Day 85 (MAD)
  PD profile of KRRO-110 based on change from Baseline in alpha-antitrypsin (AAT) enzyme levels at all measured timepoints (PiZZ participants only).
Pharmacokinetics (PK) of KRRO-110 | Day 1 to Day 43 (SAD), and Day 1 to Day 85 (MAD)
  PK profile of KRRO-110 half-life (t1/2), area under the concentration-time curve (AUC), and trough level (MAD cohorts only).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Korro Bio, Inc.
Locations (5):
- Australia (3):
  - The Prince Charles Hospital, Brisbane, Queensland
  - Nucleus Network Pty Ltd, Melbourne, Victoria
  - St. Vincent's Hospital Melbourne, Melbourne, Victoria
- New Zealand (2):
  - New Zealand Clinical Research, Auckland
  - New Zealand Clinical Research, Christchurch

IPD SHARING:
Plan to Share IPD: No